CLINICAL TRIAL: NCT00773526
Title: An Open Label Dose-escalation Study to Evaluate Safety, Pharmacokinetics and Anti-tumor Activity of RO5126766, a Dual Raf and MEK Inhibitor, Administered Orally as Monotherapy in Patients With Advanced Tumors
Brief Title: A Dose-Escalation Study of RO5126766 in Patients With Advanced Solid Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NO21895; 2008-002298-11
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — RO5126766

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: RO5126766

INTERVENTIONS:
Drug: RO5126766 — Administered orally daily for 28 days, at escalating doses (with a starting dose of 0.1mg) (Part 1). Optimal biological dose or maximum tolerated dose administered orally, daily (Part 2).

SUMMARY:
This study will determine the maximum tolerated dose and the dose limiting toxicities (Part 1 of study) and the activity (Part 2 of study) of RO5126766 in patients with metastatic or advanced solid tumors. In the first part of the study, groups of patients will by sequentially enrolled to receive ascending oral doses of RO5126766 daily for 28 days. The starting dose of 0.1mg will be escalated in subsequent groups of patients after a successful assessment of the safety and tolerability of the previous dose. In Part 2 of the study, patients with selected tumor types will be randomized to receive either the optimal biological dose or the maximum tolerated dose of RO5126766 daily. The anticipated time on study treatment is until disease progression, and the target sample size is 100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* advanced and/or metastatic cancer not amenable to standard therapy;
* any solid tumor type (Part 1); malignant melanoma, pancreatic cancer or non-small cell lung cancer (Part 2);
* measurable and/or evaluable disease (Part 1), >=1 measurable lesion (Part 2);
* ECOG performance status 0-1.

Exclusion Criteria:

* prior chemotherapy, radiotherapy or immunotherapy within 28 days of first receipt of study drug;
* prior corticosteroids as anti-cancer therapy within 14 days of first receipt of study drug;
* known past or present CNS metastases;
* acute or chronic infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (Part 1) | Throughout study
Tumor assessments (Part 2) | Event driven

SECONDARY OUTCOMES:
AEs and laboratory parameters, ophthalmological examination, pharmacokinetic parameters, pharmacodynamic parameters (Parts 1 and 2). | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Villejuif, France
- Barcelona, Barcelona, Spain
- Sutton, United Kingdom